CLINICAL TRIAL: NCT03603171
Title: Observational Trial in Myotonic Dystrophy Type 2 to Define Specific Clinical Outcome Measures
Brief Title: Clinical Outcome Measures in Myotonic Dystrophy Type 2
Acronym: COMEDY-2
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Benedikt Schoser (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Benedikt Schoser, Neurologist, senior physician, LMU Klinikum
Organization: LMU Klinikum (Other)
Other Study IDs: KlinikumUM
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Myotonic Dystrophy Type 2
Keywords: myotonic dystrophy type 2; outcome scale; muscle strength; outcome measures; disease specific severity scale
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Pain Measurement; Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM2 group: Patients with Myotonic Dystrophy type 2 genetically confirmed, without limitation regarding age or disease onset.
  Interventions: Diagnostic Test: DM1-ActivC; Diagnostic Test: R-PAct; Diagnostic Test: Beck depression inventory; Diagnostic Test: McGill pain questionnaire; Diagnostic Test: Brief Pain Inventory Short-Form; Diagnostic Test: Fatigue and Daytime Sleepiness Scale; Diagnostic Test: Myotonia Behaviour scale; Diagnostic Test: Hand opening time; Diagnostic Test: Pressure pain threshold; Diagnostic Test: Manual muscle testing; Diagnostic Test: Quantitative muscle testing; Diagnostic Test: Scale for Assessment and Rating of Ataxia; Diagnostic Test: Berg balance scale; Diagnostic Test: Quick motor function test; Diagnostic Test: GSGC; Diagnostic Test: 30 seconds sit to stand test; Diagnostic Test: Functional Index-2; Diagnostic Test: Six minute walking test; Diagnostic Test: Myotonia (from Individualised Neuromuscular Quality of Life Questionnaire)
- Healthy controls group: A group of gender and age-matched healthy controls.
  Interventions: Diagnostic Test: DM1-ActivC; Diagnostic Test: R-PAct; Diagnostic Test: Beck depression inventory; Diagnostic Test: McGill pain questionnaire; Diagnostic Test: Brief Pain Inventory Short-Form; Diagnostic Test: Fatigue and Daytime Sleepiness Scale; Diagnostic Test: Myotonia Behaviour scale; Diagnostic Test: Hand opening time; Diagnostic Test: Pressure pain threshold; Diagnostic Test: Manual muscle testing; Diagnostic Test: Quantitative muscle testing; Diagnostic Test: Scale for Assessment and Rating of Ataxia; Diagnostic Test: Berg balance scale; Diagnostic Test: Quick motor function test; Diagnostic Test: GSGC; Diagnostic Test: 30 seconds sit to stand test; Diagnostic Test: Functional Index-2; Diagnostic Test: Six minute walking test; Diagnostic Test: Myotonia (from Individualised Neuromuscular Quality of Life Questionnaire)

INTERVENTIONS:
Diagnostic Test: DM1-ActivC — A Rasch-built activity and participation scale for clinical use in myotonic dystrophy type 1 (DM1)
Diagnostic Test: R-PAct — A Rasch-built Pompe-specific activity scale.
Diagnostic Test: Beck depression inventory — A self-reported depression inventory administered verbally or self administered.
  Other Names: BDI-II
Diagnostic Test: McGill pain questionnaire — The short form of the MPQ, used to evaluate the qualitative aspect of pain and categorized in three dimensions of pain experience: sensory qualities, affective qualities and overall intensity.
  Other Names: MPQ-sf
Diagnostic Test: Brief Pain Inventory Short-Form — A 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning
  Other Names: BPI-sf
Diagnostic Test: Fatigue and Daytime Sleepiness Scale — A Rasch-built combined fatigue and daytime sleepiness scale (FDSS) specifically designed for patients with DM1.
  Other Names: FDSS
Diagnostic Test: Myotonia Behaviour scale — It consists of six framed sentences, which most closely describe the impact of the stiffness on everyday life
  Other Names: MBS
Diagnostic Test: Hand opening time — A simple test to evaluate clinical myotonia: the patient makes a tight fist for 5 seconds, then rapidly open them and the opening time is measured.
Diagnostic Test: Pressure pain threshold — Thresholds for pressure pain were obtained over eight muscles on the left and right side of the body: extensor digitorum communis, deltoid, quadriceps and anterior tibialis. The average value of two measurements will be recorded.
  Other Names: PPT
Diagnostic Test: Manual muscle testing — The patient is instructed to hold the corresponding limb or appropriate body part to be tested at the end of its available range while the practitioner provides opposing manual resistance. The strength is measured by the modified-MRC scale. The average value of two mesurements is considered. The following muscles were assessed: neck flexors and extensors, hip flexors and extensors, knee flexors and extensors, shoulder abductors, elbow flexors and extensors, ankle dorsiflexors and plantar flexors, wrist flexors and Extensors, digit flexors and extensors and thumb abductors.
  Other Names: MMT
Diagnostic Test: Quantitative muscle testing — Strength testing using sophisticated strength measuring devices during an isometric contraction. The average value of two measurements is considered; in case of difference > 10% between measurements, a third attempt is performed. The following muscles are assessed: neck flexors and extensors, hip flexors and extensors, knee flexors and extensors, shoulder abductors, elbow flexors and extensors, ankle dorsiflexors and plantar flexors, wrist flexors and extensors and digit flexors.
  Other Names: QMT
Diagnostic Test: Scale for Assessment and Rating of Ataxia — SARA is a clinical scale which assesses a range of different impairments in cerebellar ataxia.
  Other Names: SARA
Diagnostic Test: Berg balance scale — It is a 14 item objective measure designed to assess static balance and fall risk in adult populations
  Other Names: BBS
Diagnostic Test: Quick motor function test — Assessment of proximal motor function.
  Other Names: QMFT
Diagnostic Test: GSGC — GSGC score provides a detailed picture of motor function by including quantitative measures of four main motor performances (Gait, Walking, Stair, Gower's) and a qualitative global assessment of the manner to accomplish them.
Diagnostic Test: 30 seconds sit to stand test — It is a measurement that assesses functional lower extremity strenght in older adults.
  Other Names: 30CST
Diagnostic Test: Functional Index-2 — Disease-specific functional outcome assessing muscle endurance. In this trial, only the part of the test for the upper extremities is used.
  Other Names: FI-2
Diagnostic Test: Six minute walking test — It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  Other Names: 6MWT
Diagnostic Test: Myotonia (from Individualised Neuromuscular Quality of Life Questionnaire) — A subscale derived from the Individualised Neuromuscular Quality of Life Questionnaire (INQoL). 3 questions reguarding stiffness/myotonia.
  Other Names: InQoL

SUMMARY:
A monocentric, longitudinal, observational case-control study in patients with Myotonic Dystrophy type 2 (DM2). At least 60 DM2 will be evaluated through a battery of patients reported Outcomes (PROs) and clinical Outcome Measures (OMs), in order to define suitable OMs for DM2 and propose a disease specific severity scale. Patients will be re-evaluated after 6 months. An age and gender-matched control cohort will be assessed.

DETAILED DESCRIPTION:
Myotonic dystrophy type 2 (DM2) is an autosomal dominant, chronic progressive multisystemic disorder. Typical symptoms of DM2 include progressive proximal muscle weakness and wasting, often combined with axial and anterior neck muscles involvement, myotonia, muscular pain, fatigue and cataracts. The estimated prevalence is approximately 1 per 100,000 people, but in some nations as Germany the DM2 frequency is much higher than and close to 1.12.000. Compared to DM1 it has a relatively short history, as the genetic base and RNA pathogenesis have been clarified in 2003. In order to evaluate specific clinical aspects of DM2 and disease progression, the development and validation of ad-hoc tests is a unmet need in the neuromuscular field. Today, only a few outcome measures were used systematically in DM2 patients, and none of them provide so far a validation of a clinical meaningful difference for an interventional clinical trial.

The aims of this monocentric, observational, case-control study are:

1. select and validate patient reported outcomes (PRO) and outcome measures (OM) in a large group of DM2 patient
2. Propose a DM2-specific scale of disease severity
3. collecting additional information regarding the phenotype and the progression of the disease;
4. identify differences between subgroups (e.g. age, sex, years of disease).

Participants will be recruited from the German-Swiss Registry for Myotonic Dystrophy and the internal database of the Friedrich-Baur-Institute (FBI), Department of Neurology, Ludwig-Maximilian-University, Munich, Germany. A total of at least 60 male and female patients with no age limit and with genetically proven DM2 will be included. Forty age and gender-matched controls will be also assessed.

During the first evaluation of the DM2 and the controls group, the following PROs and OMs will be evaluated:

General survey (Comorbidity, BMI, familiarity, onset, etc…), DM1-ActivC, R-Pact, FDSS, McGill pain questionnaire - short form, Brief pain inventory - short form, Beck depression inventory, Myotonia behaviour scale, Myotonia subscale from INQoL, Hand opening time, pressure pain threshold, manual and quantitative muscle testing, SARA scale, Berg balance scale, QMFT, GSGC, 30 second sit and stand test, FI-2 (only for upper extremities), 6-MWT.

After six months a second evaluation of the DM2 group will be performed, in which all PROs and OMs except the general survey will be repeated.

Data analysis will provide descriptive statistic and a complete validity and reliability informations. On the basis of these results, a disease specific severity scale will be proposed for the clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed myotonic dystrophy type 2
* Able to provide informed consent

Exclusion Criteria:

* Invalidating diseases not related with DM2 (e.g. Stroke).
* Subject participating in another clinical trial (other than registries) concurrently or within 30 days prior to screening for entry into this study.
* Unable to complete study questionnaires.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Myotonic Dystrophy type 2, without limitations regarding age of onset, disease duration or physical impairment related to the disease.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Quick motor function test (QMFT) | 6 months
  A test for assessing motor function.
DM1-ActivC | 6 months
  A Rasch-built DM1 activity and participation scale for clinical use

SECONDARY OUTCOMES:
R-PAct | 6 months
  A Rasch-built Pompe-specific activity scale
Beck depression inventory (BDI-II) | 6 months
  A self-reported depression inventory administered verbally or self administered.
McGill pain questionnaire (MPQ-sf) | 6 months
  The short form of the MPQ, used to evaluate the qualitative aspect of pain and categorized in three dimensions of pain experience: sensory qualities, affective qualities and overall intensity.
Brief Pain Inventory Short-Form (BPI-sf) | 6 months
  A 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning.
Fatigue and Daytime Sleepiness Scale (FDSS) | 6 months
  A Rasch-built combined fatigue and daytime sleepiness scale (FDSS) specifically designed for patients with DM1.
Myotonia Behaviour scale (MBS) | 6 months
  It consists of six framed sentences, which most closely describe the impact of the stiffness on everyday life.
Myotonia (from Individualised Neuromuscular Quality of Life Questionnaire) | 6 months
  A subscale derived from the INQoL questionnaire. 3 questions regarding stiffness and myotonia.
Hand opening time | 6 months
  A simple test to evaluate clinical myotonia: the patient makes a tight fist for 5 seconds, then rapidly open them and the opening time is measured.
Scale for Assessment and Rating of Ataxia (SARA) | 6 months
  It is a clinical scale which assesses a range of different impairments in cerebellar ataxia.
Berg balance scale (BBS) | 6 months
  It is a 14 item objective measure designed to assess static balance and fall risk in adult populations.
Pressure pain threshold (PPT) | 6 months
  Thresholds for pressure pain were obtained over eight muscles on the left and right side of the body: extensor digitorum communis, deltoid, quadriceps and anterior tibialis. The average value oft wo measurements was recorded.
Manual muscle testing (MMT) | 6 months
  The patient is instructed to hold the corresponding limb or appropriate body part to be tested at the end of its available range while the practitioner provides opposing manual resistance. The strength is measured by the modified-MRC scale. The average value of two measurements is considered.
Quantitative muscle testing (QMT) | 6 months
  Strength testing using sophisticated strength measuring devices during an isometric contraction. The average value of two measurements is considered; in case of difference > 10% between measurements, a third attempt is performed.
GSGC | 6 months
  GSGC score provides a detailed picture of motor function by including quantitative measures of four main motor performances (Gait, Walking, Stair, Gower's) and a qualitative global assessment of the manner to accomplish them.
Functional Index-2 (only upper extremities) | 6 months
  Disease-specific functional outcome assessing muscle endurance. In this trial, only the part of the test for the upper extremities is used.
30 seconds sit to stand test (30CST) | 6 months
  It is a measurement that assesses functional lower extremity strength in older adults.
Six-minute-walking test (6MWT) | 6 months
  It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

OTHER OUTCOMES:
MIRS-2 | 10 months
  Development of a muscle impairment staging score

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Schoser, MD, Study Chair — Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen Munich, Germany
Locations (1):
- Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okkersen K, Jimenez-Moreno C, Wenninger S, Daidj F, Glennon J, Cumming S, Littleford R, Monckton DG, Lochmuller H, Catt M, Faber CG, Hapca A, Donnan PT, Gorman G, Bassez G, Schoser B, Knoop H, Treweek S, van Engelen BGM; OPTIMISTIC consortium. Cognitive behavioural therapy with optional graded exercise therapy in patients with severe fatigue with myotonic dystrophy type 1: a multicentre, single-blind, randomised trial. Lancet Neurol. 2018 Aug;17(8):671-680. doi: 10.1016/S1474-4422(18)30203-5. Epub 2018 Jun 19. PMID 29934199
- [Background] Wenninger S, Montagnese F, Schoser B. Core Clinical Phenotypes in Myotonic Dystrophies. Front Neurol. 2018 May 2;9:303. doi: 10.3389/fneur.2018.00303. eCollection 2018. PMID 29770119
- [Background] Wood L, Bassez G, van Engelen B, Lochmuller H, Schoser B; 222nd ENMC workshop participants. 222nd ENMC International Workshop:: Myotonic dystrophy, developing a European consortium for care and therapy, Naarden, The Netherlands, 1-2 July 2016. Neuromuscul Disord. 2018 May;28(5):463-469. doi: 10.1016/j.nmd.2018.02.003. Epub 2018 Feb 12. No abstract available. PMID 29550152
- [Background] Montagnese F, Mondello S, Wenninger S, Kress W, Schoser B. Assessing the influence of age and gender on the phenotype of myotonic dystrophy type 2. J Neurol. 2017 Dec;264(12):2472-2480. doi: 10.1007/s00415-017-8653-2. Epub 2017 Oct 30. PMID 29086017
- [Derived] Montagnese F, Rastelli E, Khizanishvili N, Massa R, Stahl K, Schoser B. Validation of Motor Outcome Measures in Myotonic Dystrophy Type 2. Front Neurol. 2020 Apr 21;11:306. doi: 10.3389/fneur.2020.00306. eCollection 2020. PMID 32373059